CLINICAL TRIAL: NCT04970173
Title: 1L-PEG-Asc Solution for Bowel Preparation in an "Open Access" Colonoscopy Booking System: Evaluation of Adverse Events
Status: Completed | Type: Observational
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Dr. Mauro Manno, Director, Azienda USL Modena
Other Study IDs: 01-2021
Record Dates: First submitted 2021-07-11; First posted 2021-07-21 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2021-07

CONDITIONS: Bowel Preparation
Keywords: safety
MeSH Terms: interventions — Polyethylene Glycols; MoviPrep

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: patients taking very low-volume 1L-PEG plus ascorbate (plenvu) for open access colonoscopy
  Interventions: Other: use of a very low-volume 1L-PEG plus ascorbate (plenvu) or low-volume 2L-PEG plus ascorbate (moviprep) for bowel preparation in open access colonoscopy
- 2: patients taking low-volume 2L-PEG plus ascorbate (moviprep) for open access colonoscopy
  Interventions: Other: use of a very low-volume 1L-PEG plus ascorbate (plenvu) or low-volume 2L-PEG plus ascorbate (moviprep) for bowel preparation in open access colonoscopy

INTERVENTIONS:
Other: use of a very low-volume 1L-PEG plus ascorbate (plenvu) or low-volume 2L-PEG plus ascorbate (moviprep) for bowel preparation in open access colonoscopy — Patients are free to choice the kind of BP in an open access booking system colonoscopy. The safety of BPs was assessed by reviewing the clinical and laboratory data of patients who attended the Emergency Department (ED) of the five Hospitals of our Digestive Endoscopy Unit in the 7 days following the colonoscopy. This was feasible since the electronic reporting system is the same across our five Hospitals.

SUMMARY:
Several factors are considered as the key indicators of quality colonoscopy, including endoscopist experience, withdrawal time, and quality of bowel preparation (BP). A number of laxatives are currently used as BP, and these are mainly based on PEG agents that differ for the volume and the addition of adjuvants. Several trials have demonstrated the efficacy and safety of low volume 2L-PEG based regimens compared with high volume PEG regimens and non-PEG agents. However, for low-volume 1L-PEG plus ascorbate (1L-PEG-Asc) only the data from registration trials are available, and none of these have been performed in an "open access" colonoscopy booking system. The aim of our study was to evaluate the safety and tolerability of 1L-PEG-Asc compared to 2L-PEG plus ascorbate (2L-PEG-Asc) in an "open access" booking system.

DETAILED DESCRIPTION:
All patients who underwent "open access" colonoscopy in our Unit from January 2019 to September 2020 were evaluated as part of a quality improvement project. Only patients taking 2L-PEG-Asc and 1L-PEG-Asc were enrolled in this study. Safety of BP was assessed by reviewing the number of admissions to the Emergency Department of our Hospitals and the main presentation symptom/diagnosis in the 7 days following the colonoscopy. Tolerability was evaluated as the compliance to full BP intake

ELIGIBILITY:
Inclusion Criteria:

* From January 2019 to September 2020, data from all consecutive adult (aged ≥ 18 years old) patients who underwent "open access" colonoscopy performed in our Digestive Endoscopy Unit (which is based in the Hospitals of Carpi, Castelfranco Emilia, Mirandola, Pavullo and Vignola) were collected using an electronic reporting system

Exclusion Criteria:

* Pregnant of breastfeeding patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Only consecutive patients taking Plenvu (1L-PEG-Asc, Norgine, Harefield, UK) or Moviprep (2L-PEG-Asc, Norgine, Harefield, UK) were considered in our analyses, from January 2019 to September 2020
Sampling Method: Non-Probability Sample
Enrollment: 5981 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Safety of BP was assessed by reviewing the number of admissions to the Emergency Department of our Hospitals and the main presentation symptom/diagnosis in the 7 days following the colonoscopy. | from January 2019 to September 2020
  The safety of BPs was assessed by reviewing the clinical and laboratory data of patients who attended the Emergency Department (ED) of the five Hospitals of our Digestive Endoscopy Unit in the 7 days following the colonoscopy. This was feasible since the electronic reporting system is the same across our five Hospitals.

SECONDARY OUTCOMES:
Tolerability was evaluated as the compliance to full BP intake. | from January 2019 to September 2020
  it was recorded for evert patient before the beginning of colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL Modena, Carpi, Modena, Italy

IPD SHARING:
Plan to Share IPD: No